CLINICAL TRIAL: NCT06441266
Title: Pilot Study of Multi-platform Assessment of Radiation Toxicity (M-PART) in Head and Neck Cancer Patients Treated With KeraStat® Cream for Acute Radiation Dermatitis
Brief Title: M-PART in Head and Neck Cancer Patients Treated With KeraStat Cream for Acute Radiation Dermatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00115715; P30CA012197 (NIH); ONC-HN-2404 (Other: AHWFBCCC)
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- M-PART Assessment via MyCap (Experimental): Assessment through the MyCap app to assess radiation dermatitis with the use of Kerastat cream.
  Interventions: Drug: KeraStat cream; Device: M-PART Assessments via MyCap; Other: Clinical Assessments; Other: Feedback phone interview

INTERVENTIONS:
Drug: KeraStat cream — KeraStat Cream is a non-sterile, non-implantable, emollient-based wound dressing intended to act as a protective covering in the management of a variety of skin conditions. The intervention is a topical cream applied at least twice daily starting at start of radiation therapy until 1-month from the end of radiation therapy completion
Device: M-PART Assessments via MyCap — The M-PART approach harnesses the remote data collection capabilities of MyCap to facilitate remote collection or data including but not limited to toxicity assessments, quality of life surveys, and patient-provided photographs of the skin in the treated area
Other: Clinical Assessments — Participants will undergo assessments at baseline (prior to radiation therapy start), weekly during and after radiation therapy until 1-month post-radiation therapy. Medical history will be collected at baseline including primary cancer site, HPV status (if oropharyngeal cancer primary), laterality, TNM classification, stage, surgical resection prior to radiation therapy, weight, body mass index and patient self-reported Fitzpatrick skin phototype.
Other: Feedback phone interview — Participant satisfaction, perceptions and preferences with using M-PART will be discussed.

SUMMARY:
The purpose of this research study is to test the ability of a mobile device application (MyCap) to collect patient information about their radiation skin rash in patients with head and neck cancer being treated with radiation therapy.

DETAILED DESCRIPTION:
Primary Objective: To determine the feasibility of M-PART for the assessment of acute radiation dermatitis in patients treated with radiotherapy for head and neck cancer via MyCap.

Secondary Objectives:

* To assess agreement between site clinician-rated CTCAE G2+ radiation dermatitis with moist desquamation and patient-reported moist desquamation (a and b above).
* To assess the proportion of patient-submitted photographs of skin in the irradiated area that are evaluable for radiation dermatitis assessments by central review.
* To assess agreement between clinician-rated radiation dermatitis grading, central review of patient-submitted photographs, and central review of standardized clinic photographs (methods a, c, and d above).
* To measure the level of interval (i.e., optional engagement in between scheduled collection) patient engagement in the collection of radiation toxicity outcomes using the M-PART methodology.
* To measure patient and research staff satisfaction, perceptions, and preferences with regard to the M-PART data collection framework.

OUTLINE:

Patients apply KeraStat topically at least twice daily (BID) or more as needed and complete MyCap patient reported dermatitis assessments and submit photographs in MyCap once a week (QW) during RT and for 1 month following treatment in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo clinician skin rash assessments and standardized in-clinic photography on study.

After completion of study intervention, patients may be followed for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

- Histological or cytological diagnosis of head and neck cancer (of any part of the oral cavity, pharynx, larynx, or sinuses) planned to receive conventionally fractionated radiation therapy (RT) targeting the head and neck to a total prescribed dose of at least 60 Gy. The 60 Gy RT target must include at least a part of the unilateral and/or bilateral lymph node regions of the head/neck. Planned prescribed dose will be reviewed and approved by the study PI.

NOTE: Patients without a clear pathologic diagnosis of invasive disease (i.e., biopsy showing at least carcinoma in situ) but with clinically diagnosed head and neck cancer planned for treatment as above are also eligible.

* Age ≥ 18 years at the time of enrollment.
* Able and willing to complete electronic toxicity and quality of life assessments in the MyCap application using their personal mobile device.
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative) in English.

Exclusion Criteria:

* Early stage (Stage I-II) squamous cell carcinoma of the glottic larynx planned for treatment with limited field radiation therapy alone. These participants are excluded since they are expected to receive a more limited exposure to radiation therapy.
* Patients planned for treatment to the primary site alone without regional lymph node targeting.
* Previous radiation therapy to the area in the head and neck to be treated with radiation therapy.
* Active use of topical corticosteroids in the irradiation area at the time of registration.
* History of scleroderma or active lupus requiring systemic medication at the time of registration.
* Planned concurrent treatment with anti-EGFR biologic therapy (e.g., cetuximab) for head and neck cancer.
* Individuals who are pregnant or plan to become pregnant. Radiotherapy is contraindicated in this patient population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants that Complete Scheduled Study Assessments to Measure for Feasibility | 4 weeks post radiation therapy, up to 2 years
  Participants to complete 75% or more of required assessments over the course of the study will be calculated in two steps. First, investigators will separate patients into two groups, those who have completed 75% or more of their scheduled assessments over all time periods, and those who have not. Investigators will then divide the former number by the total number of patients who completed the study (i.e., completed their radiation treatment) with a final anticipated analyzable number of 16, using a 95% confidence interval. Thus, if 50% or more of the patients in the sample have completed at least 75% of scheduled assessments, the study will be deemed feasible to conduct a future study using M-PART.

SECONDARY OUTCOMES:
Number of Participants to Self-Report Presence of Radiation Dermatitis Compared to Site Clinician Reported Radiation Dermatitis. | At baseline, weekly during radiation therapy, weekly for 4 weeks post radiation therapy, up to 2 years
  To measure agreement between site clinician reported grade 2+ radiation dermatitis with moist desquamation (yes/no) and patient-reported moist desquamation (any/none) at each weekly visit, investigators will use McNemar's test, which tests the null hypothesis that there is no difference between site clinician-reported and patient-reported presence of moist desquamation. Investigators will also estimate sensitivity and specificity (relative to the gold standard site clinician report) of the participant's self-reported moist desquamation yes/no. We will also examine whether agreement appears to vary meaningfully by week.
Percentage of Participant-Submitted Photographs Evaluable for Radiation Dermatitis Grading | At baseline, weekly during radiation therapy, weekly for 4 weeks post radiation therapy, up to 2 years
  The number of scheduled patient-submitted photographs (submitted through MyCap as part of the scheduled/required assessments) that are evaluable (if the central reviewer is able to provide a radiation dermatitis grade) in at least two different ways. First, in the most straightforward calculation, investigators will use as the denominator the total number of patient-submitted photographs that were scheduled, with the numerator being the number of photographs that are able to be graded for radiation dermatitis by a central reviewer. Second, to examine the possibility of intra-person correlation in evaluable photographs, investigators will compute for each individual patient the proportion of their photographs that were deemed evaluable and examine the distribution of these individual-level proportions in the sample. Finally, we will also carry out the above two calculations considering all photographs (scheduled and interval).
Proportion of Agreement in Grading Methods for Radiation Dermatitis | At baseline, weekly during radiation therapy, weekly for 4 weeks post radiation therapy, up to 2 years
  To assess agreement between the three different methods of grading (clinician-rated radiation dermatitis grading, participant-submitted photographs and standardized clinic photographs) investigators will compare two methods at a time in a contingency table, and estimate proportion agreeing by focusing on the diagonal where ratings of grade were identical. Investigators will also dichotomize the ordinal grades into grade 2+ yes/no and compute McNemar's test for each dichotomous comparison of ratings. Finally, investigators will also compute measures of sensitivity and specificity regarding grade 2+ yes/no again considering site clinician ratings as the gold standard.
Number of Skin Assessments Provided Through MyCap - Patient Engagement | At baseline, weekly during radiation therapy, weekly for 4 weeks post radiation therapy, up to 2 years
  To measure the level of patient engagement in the interval collection of radiation dermatitis outcomes, investigators will estimate the proportion of the total samples who provide any (vs no) interval assessment information through MyCap, and will also examine the frequency distribution of the number of such interval assessments provided among the whole sample. Additionally, investigators will make the denominator more specific by utilizing the question on the weekly scheduled patient-reported outcomes form that asks patients if they have noticed the starting or ending of moist desquamation in the interval between clinical visits, and examine what proportion of patients who answer yes on this question sent in interval information (pictures, patient-reported outcomes) during the relevant interval.
Frequency in Responses to Satisfaction with M-PART - Semi-Quantitative Survey | 4 weeks after completion of radiation therapy, up to 2 years
  The analysis of patient satisfaction, perceptions and preferences will depend on the measure of collection. For the semi-quantitative survey, investigators will compile simple descriptive statistics showing frequencies and proportions of participants in each category of response to each question.
Frequency in Responses to Satisfaction with M-PART - Qualitative Interviews | 4 weeks after completion of radiation therapy, up to 2 years
  For the qualitative interviews of patients and staff, investigators will analyze the transcripts using a thematic analysis approach. Trained qualitative researchers will review the interview transcripts and use a combined inductive-deductive approach to develop a codebook of concepts important to patient and staff satisfaction and experience with M-PART. Codes will be applied to data in a multifunctional data management and analysis software, and the codebook will be revised as needed during the analysis to best categorize and interpret the data. All transcripts will be independently coded by two researchers, and coding discrepancies will be discussed and resolved iteratively. Segments of text will be abstracted by code or groups of codes, summarized, and synthesized into themes.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan T Hughes, MD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No